CLINICAL TRIAL: NCT04935190
Title: Comparison of Resting Heart and Respiratory Rate Measurements Acquired by Contactless Radar Sensors, Electrocardiography, and Capnography
Acronym: Vitalpercept
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: DawnLight (Industry)
Responsible Party: Sponsor
Other Study IDs: CP001
Record Dates: First submitted 2021-06-14; First posted 2021-06-22 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Vital Signs

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Group 1: Subjects that have a diagnosis of a cardiac, pulmonary, or cardio-pulmonary condition (e.g., Congestive Heart Failure, COPD, Asthma) will be assigned to Group 1.
  Interventions: Diagnostic Test: Vitalpercept
- Group 2: Subjects who are not known to have a cardiac, pulmonary, or cardio-pulmonary condition will be assigned to Group 2.
  Interventions: Diagnostic Test: Vitalpercept

INTERVENTIONS:
Diagnostic Test: Vitalpercept — Comparison of resting heart and respiratory rate measurements acquired by contactless radar sensors, electrocardiography, and capnography

SUMMARY:
1. Determine agreement (accuracy) of resting heart rate measured by Vitalpercept when compared to an FDA-cleared electrocardiograph (ECG) device, LifeSignals Wireless Biosensor.
2. Determine agreement (accuracy) of resting respiratory rate measured by Vitalpercept when compared to an FDA-cleared capnographer, Capnostream 20.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects ≥ 21 years of age at the time of signing the informed consent.
2. Subjects willing to sign the informed consent and capable of committing to the duration of the study.
3. Subjects with the ability to lie flat, lie on left side, lie on right side, and sit in a chair.
4. Subjects who are able to breathe through their nose for the capnography assessment.
5. Subjects that have a diagnosis of a cardiac, pulmonary, or cardio-pulmonary condition (e.g., Congestive Heart Failure, COPD, Asthma) will be assigned to Group 1.
6. Subjects who are not known to have a cardiac, pulmonary, or cardio-pulmonary condition will be assigned to Group 2.

Exclusion Criteria:

1. Subjects who are prone to excessive coughing and excessive movement
2. Subjects who have a condition that involves uncontrollable movement of the body such as Parkinson's Disease or Essential Tremor.
3. Subjects with a history of allergy to adhesive, latex or Nuprep.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects that have a diagnosis of a cardiac, pulmonary, or cardio-pulmonary condition (e.g., Congestive Heart Failure, COPD, Asthma) will be assigned to Group 1.
  Subjects who are not known to have a cardiac, pulmonary, or cardio-pulmonary condition will be assigned to Group 2.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-06-15 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-10-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse events | During Data collection-Expected time=45-60 minutes
  Safety
Measurement of Heart Rate | During Data collection-Expected time=45-60 minutes
  Effectiveness
Measurement of Respiratory Rate | During Data collection-Expected time=45-60 minutes
  Effectiveness

CONTACTS AND LOCATIONS:
Locations (1):
- North Carolina Clinical Research, Raleigh, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No